CLINICAL TRIAL: NCT05656404
Title: Evaluation of the TorEx Lung Perfusion System in Clinical Lung Transplantation: A Safety Study
Brief Title: TorEx Lung Perfusion System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5156
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Lung Transplant; Ex Vivo Lung Perfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donor lungs assessed using TorEx Lung Perfusion System (Experimental)
  Interventions: Device: TorEx Lung Perfusion System

INTERVENTIONS:
Device: TorEx Lung Perfusion System — When donor lungs with clinical indication for EVLP are allocated to consented recipients, the lungs will be assessed using the second generation TorEx Lung Perfusion System rather than the first generation Toronto EVLP technique (standard of care).

SUMMARY:
Lung transplantation is a life-saving and life-prolonging therapy for patients with end-stage lung disease. However, the number of patients listed for lung transplantation exceeds the number of available donor lungs, leading to long wait times, deterioration in health and death of some listed patients. One way to address this issue is to reduce the number of donor lungs that are deemed unusable (declined) for transplantation. Often, donor lungs are declined for transplantation based on questionable function or inability to fully assess the organ in the donor. Due to this reason, up to 80% of potentially suitable lungs may be discarded. As a result, ex vivo lung perfusion (EVLP) was developed.

EVLP is a technique that enables the donor lungs to function in near physiological conditions outside the body, allowing surgeons to evaluate the suitability of the donor lungs for transplantation. Using this technique, centers have reported the recovery of around 70% of donor lungs that would have otherwise been deemed unusable and discarded.

The first generation Toronto EVLP technique started as a clinical trial in 2008 and became a part of the clinical standard of care at Toronto General Hospital in 2011. Since then, many clinical studies have shown that short- and long-term outcomes of recipients who received donor lungs assessed by the Toronto EVLP system were similar to those who received donor lungs deemed suitable to go straight to transplantation.

In partnership with Traferox Technologies Inc., surgeons and research team members developed the second generation TorEx Lung Perfusion System, which addresses engineering design limitations of the original Toronto EVLP system. It optimizes the Toronto EVLP technique by combining all the necessary equipment required to perform the procedure, while placing their controls within a central location. The technique of perfusion and ventilation as well as the perfusate solution remain the same between the two EVLP systems. Prior to this study, the TorEx Lung Perfusion System has not been used in clinical human lung transplantation.

The first purpose of this study is to look at the safety of using the TorEx Lung Perfusion System in 20 consented recipients. The second purpose to compare post-transplant outcomes between recipients who received donor lungs assessed by the TorEx Lung Perfusion System and a historical cohort of recipients who received donor lungs that were assessed by the first generation Toronto EVLP system.

ELIGIBILITY:
Recipient Inclusion Criteria

* Actively listed for primary lung transplantation
* Written, informed consent provided
* 18-80 years old

Recipient Exclusion Criteria

* Re-transplantation
* Multi-organ transplantation
* Participation in another interventional trial

Donor Inclusion Criteria

* Age ≤70 years old
* Ex vivo lung perfusion clinically indicated for donor lungs

Donor Exclusion Criteria

* Age >70 years old
* Donor lungs suitable to go straight to transplantation

EVLP Transplant Suitability

* Pulmonary vein PO2 > 400mmHg
* Stability or improvement of other lung function parameters during EVLP (PVR, Compliance, Airway Pressures)
* Surgeon clinically satisfied with lung evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of ISHLT Primary Graft Dysfunction Grade 3 | 72 hours post-transplant

SECONDARY OUTCOMES:
Overall survival | 30 days, 1 year post-transplant
Time on ventilator | Perioperative
ICU and hospital length of stay | Perioperative
Occurrence of acute rejection | 1 year post-transplant
Six minute walk test | 1 year post-transplant
Forced expiratory volume - one second (FEV1 in L) | 1 year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Laura Donahoe, MD MSc FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No